CLINICAL TRIAL: NCT03244085
Title: An Open-Label Phase 1b Study to Evaluate the Dose-Related Safety, Efficacy, and Pharmacokinetic Profile of Different Doses of QL-007 in Chronic Hepatitis B Patients
Brief Title: A Study to Investigate the Safety, Efficacy and Pharmacokinetic Profile of Multiple Doses of QL-007 in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QL007-002
Record Dates: First submitted 2017-07-28; First posted 2017-08-09 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100 mg BID (Experimental): Drug: QL-007 tablet; Tablet QL-007 will be administered orally daily (100 mg two times a day) over the 28 days under fasted state. Patients fast for 2h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- 200 mg BID (Experimental): Drug: QL-007 tablet; Tablet QL-007 will be administered orally daily (200 mg two times a day) over the 28 days under fasted state. Patients fast for 2h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet
- 600 mg QD (Experimental): Drug: QL-007 tablet; Tablet QL-007 will be administered orally daily (600 mg once a day) over the 28 days under fasted state. Patients fast for 2h before administration and 1h after administration.
  Interventions: Drug: QL-007 tablet

INTERVENTIONS:
Drug: QL-007 tablet — Patients will be enrolled in 1 of 3 cohorts (6 patients per cohort): QL 007 200 mg/day (100 mg BID), or QL 007 400 mg/day (200 mg/BID), or QL 007 600 mg QD. QL 007 will be administered orally daily over the 28 days under fasted state. Patients fast for 2h before administration and 1h after administration.
  Other Names: QL-007

SUMMARY:
This is a nonrandomized, open-label, no-control, dose-escalation Phase 1b trial in 18 patients with chronic HBV infection to determine the safety, preliminary efficacy, and pharmacokinetics (PK) of QL-007 after administration over 28 days of multiple oral doses in a fasted state at the following planned dose levels: 200 mg/day (100 mg two times a day (BID)), 400 mg/day (200 mg BID), then 600 mg once daily (QD), with 6 patients for each cohort.

DETAILED DESCRIPTION:
Administration of the next dose level will occur only if the preceding dose was determined to be safe and well tolerated. The decision to proceed to the next higher dose level will be made by a Safety Review Committee (SRC) based upon review of efficacy and safety data including AEs, safety laboratory results, vital signs and ECGs. PK data for up to 12 hours post-dose will also be reviewed. The review will be conducted after the last subject in a cohort completes the Day 28 visit. The planned dose levels can be modified based on the data reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 18-65 years inclusive) males or females with chronic HBV (positive for serum hepatitis B surface antigen (HBsAg) or HBV DNA for ≥ 6 months) prior to baseline.
2. Anti-HBV treatment-naive adults; adults who have taken oral anti-HBV nucleoside therapy with the last dose ≥ 4 weeks prior to screening are also eligible.
3. Positive or negative for hepatitis B e antigen (HBeAg).
4. HBV DNA ≥ 20,000 IU/mL.
5. ALT levels could be normal or elevated to < 10 times upper limit of normal.
6. Creatinine clearance ≥ 70 mL/min.
7. The following laboratory criteria have been met:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin (Hgb) ≥ 8 g/dL
   * Platelets ≥ 75 x 109/L
8. Negative serum pregnancy test for females of childbearing potential
9. For men and women who are not postmenopausal (ie, ≥ 12 months of non-therapy-induced amenorrhea, confirmed by follicle stimulating hormone (FSH), if not on hormone replacement) or surgically sterile (vasectomy in males or absence of ovaries and/or uterus or tubal ligation in females) agreement to remain abstinent or use a highly effective method of contraception during the treatment period and at least through week 12 after last dose.
10. Participants must have signed an ICF indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions.

Exclusion Criteria

Patients will be excluded from the study if one or more of the following criteria are applicable:

1. Known co-infection with HIV, hepatitis C virus (HCV) or hepatitis D virus (HDV)
2. Presence of autoimmune disorders
3. History of liver disease other than Hepatitis B
4. History of Gilbert's Disease
5. Any sign of decompensated liver disease
6. Known or suspected cirrhosis
7. Evidence of hepatocellular carcinoma
8. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

   * unstable angina within 6 months prior to screening;
   * myocardial infarction within 6 months prior to screening;
   * history of documented congestive heart failure (New York Heart Association functional classification III-IV);
   * uncontrolled hypertension defined by a systolic blood pressure (SBP) ≥ 160 mm Hg and/or diastolic blood pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication;
   * initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
   * ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication;
   * other cardiac arrhythmia not controlled with medication;
   * corrected QTc > 450 msec using Fridericia correction on the screening ECG.
9. Electrolyte abnormalities.
10. Impaired GI function or GI disease that may alter absorption of QL-007.
11. Ongoing GI AEs > grade 2 (eg, nausea, vomiting, or diarrhea) at screening.
12. Receiving medications that meet one of the following criteria and that cannot be discontinued ≥ 1 week prior to the start of treatment QL 007:

    * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (see Appendix 3; please refer to https://crediblemeds.org/pdftemp/pdf/CombinedList.pdf
    * Moderate or strong inhibitors or strong inducers of CYP3A (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Unstable or increasing doses of corticosteroids
    * Enzyme-inducing anticonvulsive agents
    * Herbal supplements.
13. Alcohol or substance abuse
14. History of bleeding diathesis
15. Patients with a history of seizures, central nervous system disorders or psychiatric disability thought to be clinically significant in the opinion of the investigator.
16. History of clinically significant gastrointestinal, cardiovascular, endocrine, renal, ocular, pulmonary, psychiatric or neurological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events of QL-007 | From randomization up to Day 36
  Safety assessments will include adverse events, clinical safety laboratory parameters, vital signs, physical examinations, and electrocardiogram results.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of QL-007 following multiple doses | On Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
The time to Cmax (tmax) of QL-007 following multiple doses | On Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
AUC0-t (area under the plasma concentration versus time curve) of QL-007 following multiple doses | On Days 1, 3, 8, 15, 22 and 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
AUC0-∞ of QL-007 following multiple doses | On Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
t1/2 (terminal elimination half-life) of QL-007 following multiple doses | On Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
Vz/F(apparent volume of distribution for the terminal disposition phase) of QL-007 following multiple doses | On Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
CL/F (apparent clearance) of QL-007 following multiple doses | On Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28, samples will be collected pre-dose; on Day 1 and 28, samples will also be collected at 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h and 12h post dose.
  Concentrations of QL-007 in plasma will be collected on Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28.
Change in serum HBsAg from baseline at Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28 | Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28
  To evaluate serum levels of HBsAg, multiple blood samples will be drawn as specified in the Schedule of Assessments. Blood samples will be collected into <[specify type of tube]> tubes during screening and on Day -1; prior to investigational product administration on Days1, 3, 8, 15, 22, 28; and on the follow-up 7 ±1 days after the last dose of the investigational product.
Change in serum HBV DNA from baseline at Day3, 8, 15, 22 and 28 | Day 1, Day 3, Day 8, Day 15, Day 22 and Day 28
  To evaluate serum levels of HBV DNA, multiple blood samples will be drawn as specified in the Schedule of Assessments. Blood samples will be collected into <[specify type of tube]> tubes during screening and on Day -1; prior to investigational product administration on Days 1, 3, 8, 15, 22, 28; and on the follow-up 7 ±1 days after the last dose of the investigational product.

CONTACTS AND LOCATIONS:
Locations (1):
- P3 Research, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided